CLINICAL TRIAL: NCT02500589
Title: Adjunctive Mood Management for Telephone-based Smoking Cessation in Primary Care
Brief Title: Adjunctive Mood Management for Telephone-based Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 11-300
Record Dates: First submitted 2015-06-24; First posted 2015-07-16 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Nicotine Dependence
Keywords: smoking; tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mood management enhancement (Experimental): In the SMK-MM enhanced arm, behavioral mood management will be integrated into the evidence-based smoking cessation counseling.
  Interventions: Behavioral: Behavioral mood management
- Health education control (Other): In the contact-equivalent health education condition, participants will receive parallel smoking cessation content on the same schedule as in the MM-enhanced arm; however, health education content will supplant the MM content. The educational content will be based on the VA National Center on Health Promotion and Disease Prevention's "Health Living Messages" on such topics as being safe, eating wisely, getting recommended immunization and screening tests, and being involved with personal health care. Participants also will receive chronic-disease-specific self-management information.
  Interventions: Other: Health education

INTERVENTIONS:
Behavioral: Behavioral mood management — The mood-management sessions are informed by CBT and emphasize psycho-educational and skills-based approaches to CBT. CBT has been used extensively to address mood management. Specifically, SMK-MM enhancement includes behavioral activation, cognitive restructuring (working with automatic thoughts, problem solving, and behavioral skills (i.e., activity scheduling, relaxation training/controlled breathing). The SMK-MM-enhanced participant manual will also include additional worksheets developed for the investigator's pilot based on Lewinsohn's self-help guide to controlling depression. The main objective of the worksheets will be to provide Veterans with an opportunity to gain mastery over selected behavioral and cognitive skills thought to facilitate mood management. As is customary in CBT, homework based on the worksheets will be discussed during counseling calls.
  Arms: Mood management enhancement
Other: Health education — In the contact-equivalent health education condition, participants will receive parallel smoking cessation content on the same schedule as in the MM-enhanced arm; however, health education content will supplant the MM content. The educational content will be based on the VA National Center on Health Promotion and Disease Prevention's "Health Living Messages" on such topics as being safe, eating wisely, getting recommended immunization and screening tests, and being involved with the participant's health care. Participants also will receive chronic-disease-specific self-management information.
  Arms: Health education control

SUMMARY:
Smoking is the leading cause of morbidity and mortality in the U.S. Interventions that increase successful quit attempts among depressed smokers with chronic medical illnesses are particularly important for the VA healthcare system because rates of tobacco use, depression, and chronic medical illnesses are significantly higher among Veterans compared to the general population. Providing smoking cessation services augmented with mood management to Veterans via telephone may increase access to, and utilization of, evidence-based smoking cessation counseling and decrease rates of smoking-related complications for Veterans with chronic medical illnesses and depression. Yet, the reach of smoking cessation telephone counseling has been limited among populations with mental illness. The investigators intend to combine the potency of co-delivered mood management and reach of telephone-delivered interventions by testing the telephone delivery of behavioral mood-management for smoking cessation among smokers with depression and chronic medical illness.

DETAILED DESCRIPTION:
Purpose: Cigarette smoking is the single greatest cause of preventable deaths. In the VA health care system, patients with chronic medical illnesses represent an important population on which to focus smoking cessation efforts. Smoking cessation among patients with chronic medical illnesses can substantially decrease morbidity and mortality. Despite these benefits, many patients with chronic medical illnesses continue to smoke. There is a strong interrelationship between depression and chronic medical illness. Depression can derail sustained smoking cessation and may be an important barrier to smoking cessation for Veterans with chronic medical illness. Despite the barriers they face, smokers with depression are motivated to quit smoking. Smokers with histories of depression may respond better to smoking cessation interventions that are augmented with mood-management adjuncts such as mood-management counseling. Thus, depressed smokers are more likely to quit when behavioral mood-management is added to traditional cessation approaches. Yet, the augmentation of smoking cessation with behavioral mood management is not yet firmly established. Also these intensive interventions have limited reach when conducted in person. Telephone counseling can deliver intensive and effective treatment to people who smoke, yet its implementation has been limited among smoker with depression. There is a need to develop novel proactive telephone-delivered approaches that can broadly deliver intensive smoking cessation interventions to Veterans who may not respond to standard care, such as those with chronic medical illnesses and depressive symptoms.

Methodology: The investigators propose a randomized comparative effectiveness trial with a two-group design in which 350 Veteran smokers with depression and chronic medical illness will be randomized to either: 1) smoking cessation plus adjunctive behavioral mood management (SMK-MM group), an intervention that includes a proactive telehealth intervention that combines evidence-based smoking cessation counseling augmented with behavioral mood management and a tele-medicine clinic for accessing nicotine replacement therapy (NRT), or 2) smoking cessation telephone counseling control (SMK CONTROL), a contact-equivalent control that provides the same smoking cessation telephone counseling intervention augmented with health education (instead of mood-management) and a tele-medicine clinic for accessing NRT. Patients with chronic medical illnesses will be identified from patient intake systems of the Durham Veteran's Affairs Hospital and screened for tobacco use and depressive symptoms.

The main outcome in this trial is prolonged abstinence at 6-month and 12-month follow-up. Logistic regression will be used to test for a between-group difference in the proportion of patients with self-reported prolonged abstinence from cigarettes at 6 months. A general linear mixed model will be used to estimate changes depressive symptoms between groups. If there is a significant intervention effect on smoking cessation, mediational analysis will be conducted to examine whether changes in self-efficacy or affect mediate the impact of the mood management intervention.

Objectives: The specific aims of the study are to 1) evaluate the impact of a telephone-delivered smoking cessation intervention augmented with behavioral mood management on rates of prolonged and point prevalence abstinence from cigarettes among Veterans with chronic medical illnesses and depression; 2) monitor the impact of behavioral mood management intervention on depressive symptoms; 3) if effective, assess whether change in self-efficacy as well as positive and negative affect mediate the impact of behavioral mood management intervention on smoking cessation among Veterans; and 4) assess the cost-effectiveness if the mood-enhanced intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria:

* 1.Enrolled in the Durham VAMC for ongoing care
* 2.Current tobacco smokers planning to quit smoking in the next 30 days
* 3.Having received a diagnosis of a qualifying chronic illness (i.e., cancer, cardiovascular disease, hypertension, diabetes, COPD)
* 4.Have significant burden of depressive symptoms (i.e., meets DSM threshold for > 3 of the nine MDD criterion symptoms at the threshold of "more than half the days" (one symptom must be depressed mood or anhedonia; endorsing "some days" meets criteria for self-harm) and endorse functional impairment OR receive a summary score 10 or above on PHQ-9.

Exclusion Criteria:

Patients who meet any one of the following exclusion criteria will be excluded:

* 1.Active diagnosis of psychosis or dementia in their medical records
* 2.Severely impaired hearing or speech
* 3.Lack of telephone access
* 4.Enrollment in another research study that might affect the main outcomes of this study
* 5.Terminal illness
* 6. Behavioral flag in medical record
* 7. Active suicidal ideation flag in medical record
* 8. Endorses thoughts of self-harm and is a greater than minimal risk of suicide

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Gierisch, PhD MA, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mood Management Enhancement | Health Education Control
Started | 175 | 175
Completed | 147 | 143
Not Completed | 28 | 32
Not completed — Withdrawal by Subject | 11 | 14
Not completed — Lost to Follow-up | 10 | 12
Not completed — Excluded post rand: cognitive impairment | 0 | 1
Not completed — Death | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Mood Management Enhancement: US veteran smokers willing to try a tobacco quit attempt with a diagnosis of a qualifying chronic illness (i.e., cancer, CVD, hypertension, diabetes, COPD), and having significant burden of depressive symptoms randomized to the mood management enhanced smoking cessation arm
- Health Education Control: US veteran smokers willing to try a tobacco quit attempt with a diagnosis of a qualifying chronic illness (i.e., cancer, CVD, hypertension, diabetes, COPD), and having significant burden of depressive symptoms randomized to the health education attention control smoking cessation arm
- Total: Total of all reporting groups
Arm/Group | Mood Management Enhancement | Health Education Control | Total
Number analyzed (Participants) | 175 | 175 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.3) | 61.8 (7.7) | 62.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 156 | 157 | 313
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 88 | 96 | 184
  White | 74 | 73 | 147
  More than one race | 8 | 1 | 9
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 175 | 175 | 350
Cigarettes per day [Count of Participants; unit: Participants] — self-report of cigarettes per day at study entry
  Participants
    10 or less | 67 | 64 | 131
    11 -20 | 76 | 77 | 153
    21-30 | 19 | 22 | 41
    31+ | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prolonged Abstinence
Description: In keeping with the Society for Research on Nicotine and Tobacco recommendations for measuring abstinence, the investigators use prolonged abstinence as the main outcome and allow for a grace period around quit date. During the 6-month follow-ups, patients will be asked about prolonged abstinence, "Since [end of the grace period] has the participant ever smoked at least a part of a cigarette on each of 7 consecutive days?" and "After [end of the grace period] has the participant smoked any in each of 2 consecutive weeks?" Responding "no" to these questions is considered having obtained prolonged abstinence (ie., smoking cessation). Data below reflect the participants responding "no."
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Mood Management Enhancement | Health Education Control
Number analyzed (Participants) | 175 | 175
Participants | 36 | 40

2. Primary Outcome: Number of Participants With Prolonged Abstinence
Description: In keeping with the Society for Research on Nicotine and Tobacco recommendations for measuring abstinence, the investigators use prolonged abstinence as the main outcome and allow for a grace period around quit date. During the 12-month follow-ups, patients will be asked about prolonged abstinence, "Since [end of the grace period] has the participant ever smoked at least a part of a cigarette on each of 7 consecutive days?" and "After [end of the grace period] has the participant smoked any in each of 2 consecutive weeks?" Responding "no" to these questions is considered having obtained prolonged abstinence (ie., smoking cessation). Data below reflect the participants responding "no."
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Mood Management Enhancement | Health Education Control
Number analyzed (Participants) | 175 | 175
Participants | 32 | 33

3. Secondary Outcome: Number of Participants With 7 Day Point Prevalent Abstinence
Description: At each follow-up (6 month), participants will be asked whether they have smoked a cigarette, even a puff, in the past 7 days and, if no, will then be asked whether the participant has smoked a cigarette, even a puff, in the past 30 days. Data presented below represents those who self-reported not smoking.
Time Frame: Month 6
Population: US veteran smokers willing to try a tobacco quit attempt with a diagnosis of a qualifying chronic illness (i.e., cancer, CVD, hypertension, diabetes, COPD), and having significant burden of depressive symptoms
Measure: Count of Participants; unit: Participants
Groups:
- Health Education Control; Mood Management Enhancement: US veteran smokers willing to try a tobacco quit attempt with a diagnosis of a qualifying chronic illness (i.e., cancer, CVD, hypertension, diabetes, COPD), and having significant burden of depressive symptoms
Arm/Group | Health Education Control | Mood Management Enhancement
Number analyzed (Participants) | 175 | 175
Participants | 37 | 35

4. Secondary Outcome: Change in PHQ-9 (Patient Depression Questionnaire) Score From Baseline to 6-months
Description: Patients were asked the frequency with which they experienced symptoms indicative of depression in the past two weeks. This measure can be used to assess Diagnostic and Statistical Manual (DSM) criterion symptoms for Major Depressive Disorder (MDD), assess depression severity, and assess suicidal ideations. The Patient Health Questionnaire-9 (PHQ-9) performs similarly across sociodemographic groups (i.e., age, race, sex) and mode of administration (e.g., patient self-report). The PHQ-9 score can range from 0 to 27, with higher scores representing higher symptom burden. We calculated the change in PHQ-9 scores from baseline to 6 month follow-up assessment. Negative scores indicate a reduction in depression symptom burden.
Time Frame: change from baseline to 6 month follow up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mood Management Enhancement | Health Education Control
Number analyzed (Participants) | 175 | 175
score on a scale | -4.53 (0.33) | -3.65 (0.34)

5. Secondary Outcome: Change in PHQ-9 (Patient Depression Questionnaire) Score From Baseline to 12 Month Follow up
Description: Patients were asked the frequency with which they experienced symptoms indicative of depression in the past two weeks. This measure can be used to assess Diagnostic and Statistical Manual (DSM) criterion symptoms for Major Depressive Disorder (MDD), assess depression severity, and assess suicidal ideations. The Patient Health Questionnaire-9 (PHQ-9) performs similarly across sociodemographic groups (i.e., age, race, sex) and mode of administration (e.g., patient self-report). The PHQ-9 score can range from 0 to 27, with higher scores representing higher symptom burden. We calculated the change in PHQ-9 scores from baseline to 12 month follow-up assessment. Negative scores indicate a reduction in depression symptom burden.
Time Frame: change from baseline to 12 month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Health Education Control | Mood Management Enhancement
Number analyzed (Participants) | 175 | 175
units on a scale | -5.09 (0.34) | -4.84 (0.35)

6. Secondary Outcome: Biochemical Verification of Smoking Cessation at 6 Month Follow up
Description: Saliva samples will be collected from participants who report not smoking in the last 7 days to biochemically validate self-report smoking status. Samples will be collected by mail within a 2-week window following the telephone interview. Data presented below represents those who were confirmed to be not smoking at 6 months via biochemical validation of of saliva samples.
Time Frame: 6 month follow up
Population: There were 23 participants who returned a sample and were not on NRT. We used a cotinine cutpoint of 15ng/mL for those not on NRT and not exposed to secondhand smoke. For those who self-reported secondhand smoke exposure, we used a cutpoint of 18ng/mL. This outcome is the number of participants whose cotinine results confirm self-report status of not smoking at the 6-month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education Control | Mood Management Enhancement
Number analyzed (Participants) | 11 | 12
Participants | 10 | 10

7. Secondary Outcome: Number of Participants With 7 Day Point Prevalent Abstinence
Description: At each follow-up (12-month), participants will be asked whether they have smoked a cigarette, even a puff, in the past 7 days and, if no, will then be asked whether the participant has smoked a cigarette, even a puff, in the past 30 days. Data presented below represents those who self-reported not smoking.
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education Control | Mood Management Enhancement
Number analyzed (Participants) | 175 | 175
Participants | 34 | 36

8. Secondary Outcome: Biochemical Verification of Smoking Cessation at 12 Month Follow up
Description: Saliva samples will be collected from participants who report not smoking in the last 7 days to biochemically validate self-report smoking status. Samples will be collected by mail within a 2-week window following the telephone interview. Data presented below represents those who were confirmed to be not smoking at 12 months via biochemical validation of of saliva samples.
Time Frame: 12 month follow up
Population: There were 32 participants who returned a sample and were not on NRT. We used a cotinine cutpoint of 15ng/mL for those not on NRT and not exposed to secondhand smoke. For those who self-reported secondhand smoke exposure, we used a cutpoint of 18ng/mL. This outcome is the number of participants whose cotinine results confirm self-report status of not smoking at the 12-month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education Control | Mood Management Enhancement
Number analyzed (Participants) | 19 | 13
Participants | 17 | 9

ADVERSE EVENTS:
Time Frame: 12 months from time of consent
Groups:
- Health Education Control: US veteran smokers willing to try a tobacco quit attempt with a diagnosis of a qualifying chronic illness (i.e., cancer, CVD, hypertension, diabetes, COPD), and having significant burden of depressive symptom
Arm/Group | Mood Management Enhancement | Health Education Control
All-Cause Mortality (participants affected / at risk) | 7/175 | 5/175
Serious Adverse Events (participants affected / at risk) | 15/175 | 15/175
Other Adverse Events (participants affected / at risk) | 82/175 | 105/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mood Management Enhancement (N=175) | Health Education Control (N=175)
Hospitlization (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hospitalization (Cardiac disorders) | 4 (4) | 3 (3)
Hospitalization (Infections and infestations) | 1 (1) | 2 (3)
Hospitalization (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Hospitalization (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hospitalization (Nervous system disorders) | 1 (1) | 1 (1)
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Hospitalization (Surgical and medical procedures) | 3 (3) | 3 (5)
Hospitalization (Vascular disorders) | 1 (1) | 1 (1)
Prolongation of Hospitalization (Infections and infestations) | 1 (1) | 0 (0)
Prolongation of Hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mood Management Enhancement (N=175) | Health Education Control (N=175)
Increased feelings of irritation, stress, or anxiety (Psychiatric disorders) | 39 (47) | 55 (88)
Flu, cold, virus, seasonal allergies, or general illness (General disorders) | 22 (23) | 21 (29)
Bodily Pain (Musculoskeletal and connective tissue disorders) | 13 (15) | 9 (32)
Craving for cigarettes (General disorders) | 8 (14) | 20 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT02500589/Prot_SAP_000.pdf